CLINICAL TRIAL: NCT03977545
Title: Assessment of Actigraphy in the Management of Neonatal Opioid Abstinence Syndrome
Brief Title: Actigraphy and Neonatal Abstinence Syndrome
Acronym: ACTINEO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018-A02290-55
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Neonatal Abstinence Syndrome
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Actigraphy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Newborn with risk of neonatal opioid abstinence syndrome (Other): The newborns will have actigraphy during 30 minutes and Lipsitz scoring system twice a day during 7 days
  Interventions: Diagnostic Test: Actigraphy
- Eutrophic term newborn (Other): The newborns will have actigraphy during 30 minutes and Lipsitz scoring system twice a day during 2 days
  Interventions: Diagnostic Test: Actigraphy
- Term newborn with low birth weight (Other): The newborns will have actigraphy during 30 minutes and Lipsitz scoring system twice a day during 2 days
  Interventions: Diagnostic Test: Actigraphy
- Eutrophic premature newborn (Other): The newborns will have actigraphy during 30 minutes and Lipsitz scoring system twice a day during 2 days
  Interventions: Diagnostic Test: Actigraphy

INTERVENTIONS:
Diagnostic Test: Actigraphy — Actigraphy will be realized twice a day during 30 minutes and Lipsitz scoring system will be realized at the same moment to analyze the correlation between Lipsitz scoring system and actigraphy in each arm.

SUMMARY:
The aim of our study is to analyse the correlation between actigraphy and Lipsitz scoring system in neonatal opioid abstinence syndrome.

DETAILED DESCRIPTION:
Neonatal opioid abstinence syndrome occurs after birth when opioids were used by the mother during pregnancy.

Many scoring systems, like Lipsitz scoring system, are used to diagnose and manage neonatal abstinence syndrome but they are subjective. The majority of items in these scores are motor skills items.

Actigraphy allows to measure objectively the newborn motricity. We will analyse the correlation between actigraphy and Lipsitz scoring system in four groups of newborns.

ELIGIBILITY:
Inclusion Criteria:

* Newborn > 32 weeks of gestation + 0 day

Exclusion Criteria:

* perinatal asphyxia
* 5- minute Apgar score < 7
* ante or post-natal brain injury diagnosis
* upper arm motor deficit
* hospitalization in intensive care unit
* neonatal respiratory distress

Max Age: 1 Day | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2019-01-23 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between actigraphy and Lipsitz scoring system | ninety minutes after feeding
  Actigraphy and Lipsitz scoring system are realized at the same time twice a day

CONTACTS AND LOCATIONS:
Locations (1):
- Caen Univerity Hospital, Caen, France